CLINICAL TRIAL: NCT04312412
Title: Outcomes of Flexor Tendons Repair in Zones I-III From 2014-2025: a Swiss Multicenter Cohort Study
Brief Title: Outcome of the Treatment of Flexor Tendon Injuries
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: BASEC-Nr. 2017-02267
Record Dates: First submitted 2020-03-04; First posted 2020-03-18 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Finger Injuries; Tendon Injury - Hand
Keywords: tendon injuries; flexor tendons
MeSH Terms: conditions — Finger Injuries; Tendon Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Controlled active motion (CAM) — Rehabilitation, post-surgery protocol

SUMMARY:
In order to gather enough data for meaningful statistics, a multicenter register of all flexor tendon repairs was established with surgical, clinical and rehabilitation patient data. The controlled active motion (CAM) protocol was administered in all patients after surgery. The purpose was to (i) measure surgery and therapy outcomes in the three centers and (ii) evaluate potential influencing factors on outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Injury between 2014 and 2025
* Flexor tendon injury of the fingers or thumb in zones 1-3

Exclusion Criteria:

* No given consent
* Concomitant injuries as fractures, large soft tissue injuries, replantation
* Bony avulsion fracture of flexor tendon (Jersey finger)
* Basic disease as rheumatoid diseases
* Primary and secondary tendon reconstruction and tendon transfer

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Range of motion | 6 weeks
  Total active motion
Range of motion | 13 weeks
  Total active motion
Range of motion | 26 weeks
  Total active motion
Range of motion | 52 weeks
  Total active motion
Grip or pinch strength | 13 weeks
  Strength
Grip or pinch strength | 26 weeks
  Strength
Grip or pinch strength | 52 weeks
  Strength
Time return to work | 52 weeks
  off work time

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Calcagni, PD Dr. med., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Clinic of Reconstructive Surgery, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beckmann-Fries V, Calcagni M, Schrepfer L, Kaempfen A, Vogelin E, Tobler-Ammann B. Relationship between pain, nerve injury and clinical outcomes after flexor tendon injuries in zones 1-2: a retrospective cohort study. Hand Ther. 2023 Jun;28(2):60-71. doi: 10.1177/17589983231159187. Epub 2023 Mar 29. PMID 37904861